CLINICAL TRIAL: NCT05137691
Title: A Feasibility RCT Investigating the Effect of a Kilocalorie Controlled, Low Carbohydrate Dietary Intervention, Behavioural Modification and Telehealth vs a Standard 1:1 NHS Weight Management Programme in Post-partum Women Living With Obesity
Brief Title: Health After Birth Intervention Trial
Acronym: HABIT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: Queen Margaret University (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Principal Investigator, Ashleigh Graham, Senior Practitioner in clinical research and Principal investigator, Queen Margaret University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10052021
Record Dates: First submitted 2021-10-18; First posted 2021-11-30 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Obesity
Keywords: weight management postpartum
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Feasibility Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Adapted NHS weight management 1:1 programme. Low carbohydrate dietary focus, enhanced behaviour change via telehealth, daily step target supported by pedometers
  Interventions: Other: Adapted NHS weight management 1:1 programme
- Active comparator NHS 1:1 weight management programme (Active Comparator): 12 week NHS 1:1 weight management programme
  Interventions: Other: NHS 1:1 weight management programme

INTERVENTIONS:
Other: Adapted NHS weight management 1:1 programme — Adapted NHS 1:1 weight management programme with a low carbohydrate dietary focus, incorporating enhanced behaviour change via telehealth, step count and pedometer
  Arms: Experimental
Other: NHS 1:1 weight management programme — NHS 1:1 weight management programme
  Arms: Active comparator NHS 1:1 weight management programme

SUMMARY:
This trial is to assess the feasibility of a larger, definitive RCT and determine the clinical effectiveness of an NHS 1:1 programme versus a modified programme with a low carbohydrate dietary intervention (as per Feinman and colleagues classification) with telehealth, physical activity and enhanced behaviour change on specified health outcomes amongst post-partum women living with obesity

DETAILED DESCRIPTION:
For individuals living with obesity, the post-partum period is currently the initial, optimal timeframe for weight management. Many women reconceive during the post-partum phase, increasing the risk of between-pregnancy bodyweight retention and even gain. Consequentially, many re-enter subsequent pregnancies with a higher BMI often associated with unfavourable obstetric outcome and further cyclical perpetuation.

Health behaviour change is an important facet within weight management interventions and delivery may be enhanced by digital technologies, for example, telehealth. Short messaging service (SMS) may be used to enhance communication between patients and practitioner and is relatively inexpensive to use.

Low carbohydrate diets continue to gain traction however research is arguably confounded by the lack of a universally agreed definition and classification. Feinman and colleagues (2015) propose intermediary categories. The experimental arm of this trial will be encouraged to adopt a non-ketogenic LCD as per Feinman.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18 or above
* Ready and motivated to make lifestyle changes
* Have a Body Mass Index of ≥30 kg/m2 (at initial booking appointment)

Additional study specific criteria

* English speaking and ability to read English language
* Capacity to consent to participating in the study
* Are non-diabetic or those with Type 2 diabetes which is diet controlled
* Deemed medically fit by GP/medical professional to participate via email
* Have recently given birth (within 1 year)
* Are not receiving weight management support elsewhere e.g. NHS, Scottish slimmers, weight watchers
* Have access to a mobile phone and weighing scales

Exclusion Criteria:

* Have uncontrolled hypothyroidism
* Have unstable psychosis or severe and unstable personality disorder
* Are pregnant
* Have dementia
* Have moderate to severe learning disability or learning difficulty which impairs the ability to adhere to the programme (identified by medical history and confirmed with GP)
* Current alcohol or substance misuse (6 month period of abstinence)
* Active purging
* Bulimia Nervosa
* Binge Eating Disorder

Additional study specific criteria

* Known cancers
* Type 1 Diabetes or Type 2 Diabetes on any Diabetic medication (including Insulin)
* Have a pacemaker
* Renal impairment
* Taking Orlistat or any other weight loss medication or had previous bariatric surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Change in Bodyweight (Kilograms) | Proposed 0,3,6,8 months
  Bodyweight measured by the CI or self-reported

SECONDARY OUTCOMES:
Change in Body composition (Fat mass/fat free mass) | Proposed 0,3,6,8 months
  Medical grade
Change in Waist circumference (Centimetres) | Proposed 0,3,6,8 months
  SECA Ergonomic measuring tape
Change in systolic and diastolic Blood pressure | Proposed 0,3,6,8 months
  Standard technique
Change in Physical activity levels | Proposed 0,3,6,8 months
  Level of physical activity (minutes) and step count from pedometer data
Change in emotional eating using the Weight loss Readiness Test II | 0,3,6,8 months
  Incidence of emotional eating (if present) determined by change score. Increased score is less favourable
Change in hunger and eating cues using the Weight loss Readiness Test II | 0,3,6,8 months
  Hunger and eating cues determined by change score. Increased score is less favourable
Change in psychological distress (if present) using the Clinical Outcomes in Routine Evaluation-10 screening tool | Baseline, post-intervention at 3 months
  Measured using the Clinical Outcomes in Routine Evaluation-10 tool using change scores. An increased score is less favourable
Change in Quality of life | Proposed 0,3,6,8 months
  Measured using the World Health Organisation Quality of life (BREF) tool. A lower score is less favourable
Food frequency questionnaire | Baseline
  Standard validated tool
Diet quality | Proposed 0,3,6,8 months
  Diet quality measured using a 3 day unweighed food diary

CONTACTS AND LOCATIONS:
Overall Officials: Ashleigh Graham, Principal Investigator — Queen Margaret University
Locations (1):
- Astley Ainslie Hospital, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only anonymised data will be accessible by the rest of the current research team for purpose of statistical analysis and monitoring